CLINICAL TRIAL: NCT01188941
Title: Linkage and Retention: A Randomized Trial to Optimize HIV/TB Care in South Africa
Acronym: Sizanani
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH); McCord Hospital (Unknown); St Mary's Hospital, London (Other); Brigham and Women's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Boston University (Other)
Responsible Party: Principal Investigator, Ingrid V. Bassett, MD, MPH, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2006-P-001379/26; R01MH090326 (NIH)
Record Dates: First submitted 2010-08-13; First posted 2010-08-26 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention)
- Assigned a Health System Navigator (Experimental)
  Interventions: Behavioral: Health System Navigator

INTERVENTIONS:
Behavioral: Health System Navigator — Subjects will be enrolled prior to an HIV test. Following TB screening, HIV infected subjects will meet with the health systems navigator who will administer a brief strengths-based interview. During this interview the participant and navigator will identify barriers to HIV and/or TB care and the resources and strengths that will be most helpful in overcoming these barriers. The health system navigator will stay in contact with participants for the next 4 months using phone calls and SMS on a standardized schedule. During the phone contacts the health system navigator will assess where the participant is on the care pathway. If the participant has not completed a step in his/her HIV or TB care, the health system navigator will help the participant draw on strengths identified in the initial interview and overcome any obstacles hindering him/her from accessing care.
  Arms: Assigned a Health System Navigator

SUMMARY:
The purpose of this study is to test the effects of a health system navigator intervention on rates of linkage to human immunodeficiency virus (HIV) and tuberculosis (TB) care among newly diagnosed HIV-infected outpatients in Durban, South Africa. Subjects will be approached in the outpatient department and enrolled prior to an HIV test. Subjects will then be randomized to the navigator arm or the standard of care arm. Subjects in the navigator arm will receive scheduled phone and short message service (SMS) contacts throughout the follow-up period to help guide them through the HIV and TB care pathways. The navigator will provide personalized support to help subjects overcome barriers they may face along the way.

DETAILED DESCRIPTION:
This project is a randomized controlled trial of an intervention to improve linkage to HIV and TB care for South Africans undergoing HIV testing. Subjects undergoing HIV testing will be enrolled at three sites in the greater Durban area. These sites comprise two hospital-affiliated outpatient departments and primary health clinics served by a mobile health van. Routine TB screening, regardless of signs or symptoms, will be offered to all HIV-infected participants. HIV-infected participants will be randomized to determine whether they will be assigned to a health system navigator or will receive the current standard of care in Durban. Block randomization will be stratified by site and gender, with blocks of varying length.

The health system navigator will help patients identify barriers to entering care and devise solutions, optimize use of available resources, and serve as a trusted social supporter who is knowledgeable about the health care system but remains outside of it. The health system navigator will help subjects engage the HIV and TB care system through face-to-face contact, telephone conversations, and short messaging service SMS text reminders which are free for patients to receive. These phone contacts and SMS will follow a standardized protocol. We will evaluate the efficacy of the intervention, as measured by increased rates of antiretroviral therapy (ART) initiation and, for those with TB co-infection, TB treatment completion. We will also evaluate the cost and cost-effectiveness of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* English or Zulu speaking
* Presenting for outpatient care
* Voluntarily undergoing an HIV test
* Able to give informed consent
* Report no prior HIV test
* Willing to share HIV and TB test results with research staff

Exclusion Criteria:

* Pregnant
* Lying in a stretcher
* Not oriented to person, place and time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1899 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Linkage and Retention in Care: ART-eligible Patients | 9 Months after Enrollment
  For ART-eligible HIV-infected patients, 3 months on ART as documented by ART initiation date in the electronic medical record.
Linkage and Retention in Care: TB Patients | 9 Months after Enrollment
  For patients co-infected with TB, 6 months of TB treatment as documented by a written discharge of treatment outcome from a TB clinic.
Linkage and Retention in Care: ART-eligible HIV/TB Co-infected Patients | 9 Months after Enrollment
  For HIV and TB co-infected patients who are ART-eligible, completion of either the ART or TB treatment outcome will be considered successful completion of the Primary Outcome Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid V Bassett, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (4):
- South Africa (4):
  - St. Mary's Hospital, Durban, KwaZulu-Natal
  - McCord Hospital, Durban, KwaZulu-Natal
  - Mariannridge Clinic, Durban, KwaZulu-Natal
  - Tshelimnyama Clinic, Durban, KwaZulu-Natal

REFERENCES:
- [Background] Bassett IV, Regan S, Chetty S, Giddy J, Uhler LM, Holst H, Ross D, Katz JN, Walensky RP, Freedberg KA, Losina E. Who starts antiretroviral therapy in Durban, South Africa?... not everyone who should. AIDS. 2010 Jan;24 Suppl 1(Suppl 1):S37-44. doi: 10.1097/01.aids.0000366081.91192.1c. PMID 20023438
- [Background] Losina E, Bassett IV, Giddy J, Chetty S, Regan S, Walensky RP, Ross D, Scott CA, Uhler LM, Katz JN, Holst H, Freedberg KA. The "ART" of linkage: pre-treatment loss to care after HIV diagnosis at two PEPFAR sites in Durban, South Africa. PLoS One. 2010 Mar 4;5(3):e9538. doi: 10.1371/journal.pone.0009538. PMID 20209059
- [Background] Drain PK, Losina E, Parker G, Giddy J, Ross D, Katz JN, Coleman SM, Bogart LM, Freedberg KA, Walensky RP, Bassett IV. Risk factors for late-stage HIV disease presentation at initial HIV diagnosis in Durban, South Africa. PLoS One. 2013;8(1):e55305. doi: 10.1371/journal.pone.0055305. Epub 2013 Jan 28. PMID 23383147
- [Background] Regan S, Losina E, Chetty S, Giddy J, Walensky RP, Ross D, Holst H, Katz JN, Freedberg KA, Bassett IV. Factors associated with self-reported repeat HIV testing after a negative result in Durban, South Africa. PLoS One. 2013 Apr 23;8(4):e62362. doi: 10.1371/journal.pone.0062362. Print 2013. PMID 23626808
- [Background] Bassett IV, Giddy J, Chaisson CE, Ross D, Bogart LM, Coleman SM, Govender T, Robine M, Erlwanger A, Freedberg KA, Katz JN, Walensky RP, Losina E. A randomized trial to optimize HIV/TB care in South Africa: design of the Sizanani trial. BMC Infect Dis. 2013 Aug 26;13:390. doi: 10.1186/1471-2334-13-390. PMID 23972276
- [Background] Drain PK, Losina E, Coleman SM, Giddy J, Ross D, Katz JN, Bassett IV. Rapid urine lipoarabinomannan assay as a clinic-based screening test for active tuberculosis at HIV diagnosis. BMC Pulm Med. 2016 Nov 14;16(1):147. doi: 10.1186/s12890-016-0316-z. PMID 27842535
- [Background] Bassett IV, Coleman SM, Giddy J, Bogart LM, Chaisson CE, Ross D, Flash MJ, Govender T, Walensky RP, Freedberg KA, Losina E. Barriers to Care and 1-Year Mortality Among Newly Diagnosed HIV-Infected People in Durban, South Africa. J Acquir Immune Defic Syndr. 2017 Apr 1;74(4):432-438. doi: 10.1097/QAI.0000000000001277. PMID 28060226
- [Background] Drain PK, Losina E, Coleman SM, Bogart L, Giddy J, Ross D, Katz JN, Bassett IV. Social support and mental health among adults prior to HIV counseling and testing in Durban, South Africa. AIDS Care. 2015;27(10):1231-40. doi: 10.1080/09540121.2015.1046417. Epub 2015 Jul 25. PMID 26213142
- [Background] Drain PK, Losina E, Coleman SM, Giddy J, Ross D, Katz JN, Bassett IV. Value of urine lipoarabinomannan grade and second test for optimizing clinic-based screening for HIV-associated pulmonary tuberculosis. J Acquir Immune Defic Syndr. 2015 Mar 1;68(3):274-80. doi: 10.1097/QAI.0000000000000436. PMID 25415288
- [Background] Drain PK, Losina E, Coleman SM, Giddy J, Ross D, Katz JN, Walensky RP, Freedberg KA, Bassett IV. Diagnostic accuracy of a point-of-care urine test for tuberculosis screening among newly-diagnosed HIV-infected adults: a prospective, clinic-based study. BMC Infect Dis. 2014 Feb 26;14:110. doi: 10.1186/1471-2334-14-110. PMID 24571362
- [Background] Cohen GM, Drain PK, Noubary F, Cloete C, Bassett IV. Diagnostic delays and clinical decision making with centralized Xpert MTB/RIF testing in Durban, South Africa. J Acquir Immune Defic Syndr. 2014 Nov 1;67(3):e88-93. doi: 10.1097/QAI.0000000000000309. PMID 25314255
- [Result] Bassett IV, Coleman SM, Giddy J, Bogart LM, Chaisson CE, Ross D, Jacobsen MM, Robine M, Govender T, Freedberg KA, Katz JN, Walensky RP, Losina E. Sizanani: A Randomized Trial of Health System Navigators to Improve Linkage to HIV and TB Care in South Africa. J Acquir Immune Defic Syndr. 2016 Oct 1;73(2):154-60. doi: 10.1097/QAI.0000000000001025. PMID 27632145
- [Derived] Bassett IV, Xu A, Giddy J, Bogart LM, Boulle A, Millham L, Losina E, Parker RA. Changing contextual factors from baseline to 9-months post-HIV diagnosis predict 5-year mortality in Durban, South Africa. AIDS Care. 2021 Dec;33(12):1543-1550. doi: 10.1080/09540121.2020.1837338. Epub 2020 Nov 2. PMID 33138630
- [Derived] Platt L, Xu A, Giddy J, Bogart LM, Boulle A, Parker RA, Losina E, Bassett IV. Identifying and predicting longitudinal trajectories of care for people newly diagnosed with HIV in South Africa. PLoS One. 2020 Sep 21;15(9):e0238975. doi: 10.1371/journal.pone.0238975. eCollection 2020. PMID 32956380
- [Derived] Bajema KL, Bassett IV, Coleman SM, Ross D, Freedberg KA, Wald A, Drain PK. Subclinical tuberculosis among adults with HIV: clinical features and outcomes in a South African cohort. BMC Infect Dis. 2019 Jan 5;19(1):14. doi: 10.1186/s12879-018-3614-7. PMID 30611192